CLINICAL TRIAL: NCT02358109
Title: Cost-Effectiveness of an Exercise Program in Midlife Women
Brief Title: The Flamenco (Fitness League Against MENopause COsts) Project
Acronym: FLAMENCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Collaborators: Andalusian Regional Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Virginia A. Aparicio García-Molina, PhD Sport Sciences, PhD Nutrition and Food Technology, Universidad de Granada
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: FLAMENCO
Record Dates: First submitted 2014-09-23; First posted 2015-02-06 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Cardiovascular Diseases; Diabetes; Dyslipidemias; Metabolic Syndrome; Quality of Life
Keywords: Cost-Benefit Analysis, Exercise,Women,Diseases/Prevention
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Dyslipidemias; Metabolic Syndrome; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention arm (Experimental): Intervention group receive directed classes of physical conditioning, 3 hours/week during a period of 16 weeks
  Interventions: Behavioral: exercise
- Control arm (No Intervention): Control group do not receive physical conditioning intervention but usual care advice and are measured at the beginning and at the end of the study

INTERVENTIONS:
Behavioral: exercise — The exercise intervention will be performed in groups of 20 participants which will train 3 days/week (60 min per session) for a 16-week period. Sessions will be designed and carefully supervised by exercise monitors, including a 15 minute warm-up period followed by 35 minute focused on aerobic exercises, developed progressively at intensity sufficient to achieve 50% (at the beginning of the intervention) and 80% (the last month of the intervention) of predicted maximum heart rate (209-0.73 × age) and resistance strength training.Monday sessions will involve resistance strength exercises. Wednesday sessions will include balance oriented activities and dancing aerobic exercises. Fridays will include aerobic, resistance strength and coordination using a circuit of different exercises.Sessions finish with a 10 minute cool-down period of stretching and relaxation exercises.
  Arms: Intervention arm

SUMMARY:
Spain is the second country in the world that consume more drugs. The average drug expenditure per capita in Andalucía during 2011 was 219.2 €. This drug spending increases during the perimenopausal period. According to the Study of the Economic Impact of Sport on Health Spending of the Ministry of Health of the Generalitat of Catalonia, for every euro invested in sports promotion 50 euros are saved in health spending accumulated over 15 years. The main objectives of this project are: i) To analyze the (cost-effectiveness) effect of an exercise program on the prescription of drugs in a sample of Andalusian women aged 45-60 years. ii ) To study the level of physical activity and sedentarism (measured objectively by accelerometry ) , functional capacity , quality of life and clinical profile of this population. iii ) To analyze the relationship between levels of physical activity / sedentarism and pharmaceutical expenditure. In the present project, an exercise program aimed at minimizing symptoms and health problems associated with the perimenopausal period will be performed (Dyslipidemia, diabetes, anxiety, depression, quality of life, quality of sleep, obesity, osteoporosis and cardiovascular disease). A total of 160 perimenopausal women will be randomly assigned to the intervention group exercise (n = 80 ) or to the usual care group (n = 80). Participants in the intervention group will train 3 days / week ( 60 min per session ) for 16 weeks.

With the analysis of the results of this project new patterns of objective work as well as the most significant practical resources for the design of a master plan may be determined. Results are expected to be able to shed some light on the implementation of programs of health promotion that are both time beneficial for the Andalusian Public Health and for the family , institutional and community economy.

DETAILED DESCRIPTION:
Spain is the second country in the world that consumes more drugs. The average drug expenditure per capita in Andalucía during 2011 was 219.2 €. This drug spending increases during the perimenopausal period. According to the Study of the Economic Impact of Sport on Health Spending of the Ministry of Health of the Generalitat of Catalonia, for every euro invested in sports promotion 50 euros are saved in health spending accumulated over 15 years. The main objectives of this project are: i) To analyze the (cost-effectiveness) effect of an exercise program on the prescription of drugs in a sample of Andalusian women aged 45-60 years. ii ) To study the level of physical activity and sedentarism (measured objectively by accelerometry ) , functional capacity , quality of life and clinical profile of this population. iii ) To analyze the relationship between levels of physical activity / sedentarism and pharmaceutical expenditure. In the present project, an exercise program aimed at minimizing symptoms and health problems associated with the perimenopausal period will be performed (Dyslipidemia, diabetes, anxiety, depression, quality of life, quality of sleep, obesity, osteoporosis and cardiovascular disease). A total of 160 perimenopausal women will be randomly assigned to the intervention group exercise (n = 80 ) or to the usual care group (n = 80). Participants in the intervention group will train 3 days / week ( 60 min per session ) for 16 weeks.

With the analysis of the results of this project new patterns of objective work as well as the most significant practical resources for the design of a master plan may be determined. Results are expected to be able to shed some light on the implementation of programs of health promotion that are both time beneficial for the Andalusian Public Health and for the family , institutional and community economy.

The present study is a Randomized Controlled Trial (RCT). The study protocols were approved by the Ethics Committee for Research Involving Human Subjects at the University of Granada. All participants have to provide a written informed consent. After baseline measurements, they will be randomly allocated to the usual care (control) or exercise intervention group. The participants will be followed for 16 weeks during the training interventions. All the baseline and follow-up examinations will be performed in the same setting (two primary care health centers) and by the same researchers. The study will follow the ethical guidelines of the Declaration of Helsinki (last modified in 2013).

Participants at the control group will receive general advices about the positive effects of physical activity by pamphlets describing the benefits their benefits and general guidelines about how to increase the daily physical activity levels.

The exercise intervention will be performed in groups of 20 participants. Each group will train 3 days/week (60 min per session) for a 16-week period. It will meet the minimum training standards of the American College of Sports Medicine(Garber, Blissmer et al. 2011). Each exercise session will be designed and supervised by exercise monitors and will include a 15 minute warm-up period followed by 35 minute focused mainly on aerobic exercises, developed progressively and resistance strength training.

Monday sessions will involve resistance strength exercises developed at a slow pace including a stepped progression during the program. Resistance strength training will include 1-3 set of 12-20 repetitions of 8-10 exercises involving all major muscle groups. The strengthening exercises will include biceps curls, arm extensions, arm side lifts, shoulder elevations, lateral leg elevations, stands up from seated position, lunge, sideways lunge and step-up/step-down and similar exercises. The load will be gradually increased as the strength of each person improves. Body weight and barbells will be used at the start of the program. Wednesday sessions will include balance oriented activities and dancing aerobic exercises. Fridays will include aerobic, resistance strength and coordination using a circuit of different exercises. The exercise sessions will finish with a 10 minute cool-down period of stretching and relaxation exercises.

Heart rate will be assessed with a heart rate monitor (Polar Electro OY, Finland) in order to control the intensity of the sessions. One third of the patients in the intervention group will wear heart rate monitors in 1/3 of the sessions, randomly selected. The rate of perceived exertion (RPE) will be monitored using the Borg's conventional (6-20 point) scale(Borg 1982). Intensity (expressed as RPE) will range from 12 to 16-17. To maximize adherence, several strategies will be implemented including music in all sessions, individualized attention at the intervention sessions and telephone calls following missed sessions. Make-up sessions will be allowed in case of missing sessions (due to illness or any other reason).

During the Flamenco Project development X main measurement categories will be assessed: 1) socio-demographic and clinical information; 2) blood pressure and resting heart rate; 3) body composition; 4) physical fitness; 5) physical activity and sedentary behaviour; 6) sleep quality; 7) fatigue; 8) mental health; 9) dietary patterns and 10) hormonal, glycemic and lipid profile.

First, the participants will be cited for the blood analysis. Secondly, they will have to attend to the primary care health center for the socio-demographic and clinical information, blood samples extraction, blood pressure and resting heart rate, body composition and physical fitness assessments. This day, the participant will receive the accelerometer and nine days later she will have to return it in the same primary care health center. During those nine days, the participants will have to complete the questionnaires

1. Socio-demographic and clinical information will be collected using a questionnaire regarding smoking and alcohol habits, history of illness, menopause status and symptoms, indicators of socio-economic status, marital status and number of children. The pharmacology registry will be consulted by the primary health care staff in the medical database.
2. Blood pressure and resting heart rate, systolic and diastolic blood pressure, as well as resting heart rate, will be measured after 5 minutes of rest, two times with 2 minutes apart, with the participant seated. The lowest value will be selected for the analysis.
3. Body Composition: Lean, fat and bone mass of the whole body will be measured. Height (cm) and waist circumference (cm) will be also assessed.
4. Physical fitness will be assessed by means of the following tests:

   * Lower body muscular strength: The "30-s chair stand test" involves counting the number of times within 30 s that an individual can rise to a full stand from a seated position with back straight and feet flat on the floor, without pushing off with the arms(Rikli and Jones 1999).
   * Upper body muscular strength: The "Arm curl test" involves determining a number of times a hand weight (2.3 kg for women) can be curled through a full range of motion in 30 s. Additionally, handgrip strength will be measured using a digital dynamometer (TKK 5101 Grip-D; Takey, Tokyo, Japan) (Ruiz-Ruiz, Mesa et al. 2002).
   * Lower body flexibility: It will be used the Sit and Reach test(Rodriguez, Gusi et al. 1998) and an adaptation of it called the "Back Saver Sit and Reach" test
   * Upper body flexibility by the "back scratch test", a measure of overall shoulder range of motion(Rikli and Jones 1999).
   * Motor agility: timed up and go test(Podsiadlo and Richardson 1991).
   * Static balance: It was assessed with the Blind Flamingo test(Rodriguez, Gusi et al. 1998) with eyes closed.
   * Cardiorespiratory fitness: The modified Bruce protocol(Bruce, Kusumi et al. 1973; Gulati, Pandey et al. 2003) will be performed to estimate maximal oxygen uptake (VO2max), which will be used as measure of cardiorespiratory fitness in the present study. Additionally, the "6-min walk " test(Rikli and Jones 1999) will be evaluated. This test involves determining the maximum distance (meters) that can be walked in 6 min along a 45.7 m rectangular course.
5. Physical activity and sedentary behaviour will be subjectively and objectively assessed:

   * Accelerometry: Participants will be asked to wear a tri-axial accelerometer (ActiGraph GT3X+, Pensacola, Florida, US) for 9 consecutive days, starting the same day the monitor was received. Participants will be instructed on how to wear it.
   * The Leisure Time Physical Activity Instrument, the Physical Activity at Homework or Workplace Instrument (Mannerkorpi and Hernelid 2005; Munguia-Izquierdo, Legaz-Arrese et al. 2011), the Spanish version of the Sedentary Behaviour Questionnaire(Rosenberg, Norman et al. 2010; Munguia-Izquierdo, Segura-Jimenez et al. 2013) and the short version of the ALPHA Environmental questionnaire(Spittaels, Foster et al. 2009; Spittaels, Verloigne et al. 2010).
6. Sleep quality will be assessed by the Pittsburgh Sleep Quality Index(Buysse, Reynolds et al. 1989), which assesses sleep quality and disturbances over a l-month time interval.
7. Fatigue will be assessed by The Multidimensional Fatigue Inventory-Spanish(Munguia-Izquierdo, Segura-Jimenez et al. 2012) which is a 20-item assessment tool with five domains: general fatigue, physical fatigue, mental fatigue, reduced activity, and reduced motivation.
8. Mental Health will be evaluated by a wide range of tests: Mini Mental State Examination(Folstein, Folstein et al. 1975), the Short-Form Health Survey 36 (SF-36) (Alonso, Prieto et al. 1995), the Spanish version of the Rosenberg Self-Esteem Scale(Vazquez, Jimenez et al. 2004), the Subjective Happiness Scale(Lyubomirsky and Lepper 1999; Extremera and Fernández-Berrocal 2013), the 10-item Connor-Davidson Resilience Scale(Campbell-Sills and Stein 2007; Notario-Pacheco, Solera-Martinez et al. 2011), the brief COPE(Carver 1997; Morán, Landero et al. 2009), the Beck Depression Inventory-II(Beck, Ward et al. 1961; Beck, Steer et al. 2006), the State Trait Anxiety Inventory (Spielberger CD, Gorsuch RL et al. 2002); mood state will be assessed using a Profile of Mood State questionnaireMcNair D.M., Lorr M., Droppleman L.F. Revised Manual for the Profile of Mood States. Educational and Industrial Testing Services; San Diego, CA, USA: 1992.

   Positive health will be assessed by means of the following questionnaires: the Trait Meta-Mood Scale(Fernandez-Berrocal, Extremera et al. 2004), the Positive and Negative Affectivity Schedule(Watson, Clark et al. 1988; Sandín, Chorot et al. 1999), the Satisfaction With Life Scale(Diener, Emmons et al. 1985; Atienza, Pons et al. 2000) and the Life Orientation Test Revised(Scheier, Carver et al. 1994; Otero, Luengo et al. 1998) The EuroQol 5D (EQ-5D) will be used to assess five dimensions of health related quality of life: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, each of which is defined through five severity levels(Badia, Roset et al. 1999; Herdman, Badia et al. 2001).
9. Dietary patterns will be evaluated by the Food Frequency Questionnaire and the Mediterranean Diet Score created by Panagiotakos et al. in 2006(Panagiotakos, Pitsavos et al. 2006)
10. Hormonal, glycemic and lipid profile will be assess by the blood sample collection with standard methods using an autoanalyzer.

The analysis in this study will be a cost-utility analysis with a health system perspective. It will be conducted considering the costs and the health effects of the intervention. The measurement of health effects will be the Quality Adjusted Life Years (QALYs).

This study try to determine the effectiveness and cost-effectiveness of a primary health care-based exercise intervention aimed to reduce CVD risk, improve body composition, physical fitness and mental health in middle-aged women.

ELIGIBILITY:
Inclusion Criteria:

* Age: 45-60 years.
* Not to have other severe somatic or psychiatric disorders, or other diseases that prevent physical loading (Answer "no" to all questions on the Physical Activity Readiness Questionnaire-PAR-Q) .
* Not to be engaged in regular physical activity >20 min on >3 days/week.
* Able to ambulate, with or without assistance.
* Able to communicate.
* Informed consent: Must be capable and willing to provide consent.

Exclusion Criteria:

* Acute or terminal illness.
* Myocardial infarction in the past 3 months.
* Not capable to ambulate.
* Unstable cardiovascular disease or other medical condition.
* Upper or lower extremity fracture in the past 3 months.
* Severe dementia (MMSE < 10).
* Unwillingness to either complete the study requirements or to be randomised into control or training group.
* Presence of neuromuscular disease or drugs affecting neuromuscular function.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2014-01; Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The Incremental Cost Effectiveness Ratio (ICER) | 16 weeks
  It is calculated dividing the difference between the average costs of both groups by the difference in mean QALYs gained in both groups.

SECONDARY OUTCOMES:
Quality Adjusted Life Years (QALYs) | 16 weeks
  This is an average of cost and effectiveness (the mean QALYs gained) in both groups, control and intervention. The QALYs are calculated multiplying the years of life by the patient's quality of life. The Patients' quality of life will be assessed by the EQ-5D questionnaire.

OTHER OUTCOMES:
Blood pressure | 16 weeks
  Systolic and diastolic blood pressure will be measured after 5 minutes of rest, two times 2 minutes apart, with the person sit down (Omron Health Care Europe B.V. Hoolddorp). The lowest value of two trials will be selected for the analysis.
Resting heart rate | 16 weeks
  Resting heart rate will be measured after 5 minutes of rest, two times 2 minutes apart, with the person sit down (Omron Health Care Europe B.V. Hoolddorp). The lowest value of two trials will be selected for the analysis.
Body composition | 16 weeks
  Lean, fat and bone mass of the whole body will be measured using dual-energy x-ray absorptiometry (DXA) with a Hologic QDR-4500A device (software version 11.2.1; Hologic, Bedford, MA, USA). Height (cm) will be measured using a stadiometer (Seca 22, Hamburg, Germany). Waist circumference (cm) will be assessed with the participant standing at the middle point between the ribs and the ileac crest (Harpenden anthropometric tape, Holtain Ltd).
Lower body muscular strength | 16 weeks
  The "30-s chair stand" test involves counting the number of times within 30 s that an individual can rise to a full stand from a seated position with back straight and feet flat on the floor, without pushing off with the arms. The patients will perform one trial after familiarization
Upper body muscular strength | 16 weeks
  The "Arm curl" test involves determining a number of times a hand weight (2.3 kg for women) can be curled through a full range of motion in 30 s. Additionally, handgrip strength will be measured using a digital dynamometer (TKK 5101 Grip-D;Takey, Tokyo, Japan) as described elsewhere. Patients will perform (alternately with both hands) the test twice allowing a 1-min rest period between measures. The best value of 2 trials for each hand will be chosen and the average of both hands will be used in the analyses.
Lower body flexibility | 16 weeks
  The "Sit and Reach" test in which participant will be required to sit with knees straight and legs together, and feet placed against the box. The participant slowly reached forward as far as possible. The final position that the participant reached in centimeters will be the score for the test. The best score of two attempts will be recorded.
Upper body flexibility | 16 weeks
  The "back scratch" test, a measure of overall shoulder range of motion, involves measuring the distance between (or overlap of) the middle fingers behind the back with a ruler. Participants will perform this test twice, alternately with both hands, and the best value will be registered. The average of both hands will be used in the analyses.
Motor agility/dynamic balance | 16 weeks
  "Timed up and go test",with the participant sit in a chair (seat height 44 cm, depth 45 cm, width 49 cm, armrest height 64 cm) with arms and trunk supported. Subjects will be instructed to stand up on the word "go" and walk three meters in a straight line, turned 180 degrees, walk back to the chair and sit down again in the chair. Each subject will perform 1 trial to become familiar with the test. After a 1-minute rest, the test will be performed twice separated by a 1-minute rest. The time from the start until the subject sit down in the chair with back support will be measured and the better of the 2 attempts will be used in the data analysis.
Static balance | 16 weeks
  It will be assessed through the blind flamingo test with closed eyes. In this test, the number of trials needed to complete 30 s of the static position is recorded, and the chronometer is stopped whenever the patient does not comply with the protocol conditions. One trial will be accomplished for each leg and the average of both values will be selected for the analysis.
Cardiorespiratory fitness | 16 weeks
  The modified Bruce protocol will be used as measure of cardiorespiratory fitness The test consists of 5 increasing workload stages of 3 minutes each (stage 1: 1.7mph and 10% inclination; stage 2: 2.5mph and 12% inclination; stage 3: 3.4mph and 14% inclination; stage 4: 4.2mph and 16% inclination; stage 5: 5mph and 18% inclination). The test will terminate when the 85% of the individual's heart rate reserve (HRR) will be accomplished. VO2max will be estimated with the formula by Bruce et al.: VO2max= 6.70 - 2.82*2 + 0.056*duration of the test. Additionally, we will also assess the "6-minutes walk" test. This test involves determining the maximum distance (meters) that can be walked in 6 minutes along a 45.7 m rectangular course.
Physical activity | 16 weeks
  It will be used a tri-axial accelerometer (ActiGraph GT3X+, Pensacola, Florida, US) for 8 consecutive days. Monitor wearing time will be calculated by subtracting the non-wear time and the sleeping time (recorded through a diary) from the total registered time for the entire day. A total of 7 days of recording with a minimum of ten or more hours of registration per day will be necessary to be included in the study. Physical activity levels will expressed as mean counts per minute. This is a measure of overall physical activity. We will calculate mean counts per minute by dividing the sum of total counts per epoch for a valid day by the number of minutes of wear time in that day across all valid days. We will also calculate the time engaged in light, lifestyle, moderate, and moderate and vigorous intensity physical activity based upon a standardized cut-offs.
Sedentary behaviour | 16 weeks
  It will be used a tri-axial accelerometer (ActiGraph GT3X+, Pensacola, Florida, US) for 8 consecutive days. Monitor wearing time will be calculated by subtracting the non-wear time and the sleeping time (recorded through a diary) from the total registered time for the entire day. A total of 7 days of recording with a minimum of ten or more hours of registration per day will be necessary to be included in the study. Sedentary time will be calculated as the amount of time accumulated below 100 counts per minute during periods of wear time.
Sleep Quality | 16 weeks
  The Pittsburgh Sleep Quality Index will be used to assess sleep quality and disturbances over a l-month time interval. Nineteen individual items generate seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score.
Fatigue | 16 weeks
  The Multidimensional Fatigue Inventory-Spanish is a 20-item assessment tool with five domains: General Fatigue, Physical Fatigue, Mental Fatigue, Reduced Activity, and Reduced Motivation. Each domain consists of four items and has a potential score range from 4 to 20, where higher scores indicate a high degree of fatigue.
Mediterranean Diet Score (MDS) | 16 weeks
  It evaluates the degree of adherence to the traditional Mediterranean dietary pattern. It consists on 11 items and scores ranging from 0-5 based on frequency of consumption (servings/month: Never, 1-4, 5-8, 9-12, 13-18, >18). Seven of them scores positively with increased consumption, as they are components of the Mediterranean Diet (non-refined cereals, potatoes, fruits, vegetables, legumes, fish, and olive oil). The score of the item "use of olive oil" in cooking ranges from never (0) to daily (5) (times/week). Red meat and derivates, poultry and full fat dairy products score positively with less consumption. Especially for alcohol, the score 5 is assigned for consumption of less than 300 ml/day, score 0 for consumption of more than 700 ml/day or none and scores 1-4 for consumption of 300-400, 400-500, 500-600, and 600-700 ml/day, respectively. Thus, the total score assigned ranges from 0-55, with higher scores indicating greater adhesion to the Mediterranean diet pattern.
Hemogram profile | 16 weeks
  Venous blood samples will be taken in vacuum tubes in standardized fasting conditions at 8-9 am in the primary care health center and transported to the laboratory for their posterior analysis. Two vacuum tubes will be collected for each participant and one of them will contain EDTA/K3 to determine blood cells count, blood hemoglobin concentration and hematocrit. Plasma total cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol, triglycerides, glucose, insulin, albumin, total proteins, creatinine, uric acid, creatine kinase, sodium, potassium, glycosylated hemoglobin and thyroid-stimulating hormone levels will be assessed with standard methods using an autoanalyzer (Hitachi-Roche p800, F. Hoffmann-La Roche Ltd. Switzerland).

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Aparicio García-Molina, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Department of Physiology, Faculty of Farmacy, University of Granada, Granada, Andalusia, Spain

REFERENCES:
- [Background] Gulati M, Pandey DK, Arnsdorf MF, Lauderdale DS, Thisted RA, Wicklund RH, Al-Hani AJ, Black HR. Exercise capacity and the risk of death in women: the St James Women Take Heart Project. Circulation. 2003 Sep 30;108(13):1554-9. doi: 10.1161/01.CIR.0000091080.57509.E9. Epub 2003 Sep 15. PMID 12975254
- [Background] Mannerkorpi K, Hernelid C. Leisure Time Physical Activity Instrument and Physical Activity at Home and Work Instrument. Development, face validity, construct validity and test-retest reliability for subjects with fibromyalgia. Disabil Rehabil. 2005 Jun 17;27(12):695-701. doi: 10.1080/09638280400009063. PMID 16012062
- [Background] Otero, J. M., A. Luengo, et al. (1998). Psicología de la Personalidad. Manual de prácticas. Barcelona, Ariel Practicum.
- [Background] Sandín, B., P. Chorot, et al. (1999).
- [Background] Scheier MF, Carver CS, Bridges MW. Distinguishing optimism from neuroticism (and trait anxiety, self-mastery, and self-esteem): a reevaluation of the Life Orientation Test. J Pers Soc Psychol. 1994 Dec;67(6):1063-78. doi: 10.1037//0022-3514.67.6.1063. PMID 7815302
- [Background] Extremera, N. and P. Fernández-Berrocal (2013).
- [Result] Alonso J, Prieto L, Anto JM. [The Spanish version of the SF-36 Health Survey (the SF-36 health questionnaire): an instrument for measuring clinical results]. Med Clin (Barc). 1995 May 27;104(20):771-6. Spanish. PMID 7783470
- [Result] Pons D, Atienza FL, Balaguer I, Garcia-Merita ML. Satisfaction with life scale: analysis of factorial invariance for adolescents and elderly persons. Percept Mot Skills. 2000 Aug;91(1):62-8. doi: 10.2466/pms.2000.91.1.62. PMID 11011872
- [Result] Badia X, Roset M, Montserrat S, Herdman M, Segura A. [The Spanish version of EuroQol: a description and its applications. European Quality of Life scale]. Med Clin (Barc). 1999;112 Suppl 1:79-85. Spanish. PMID 10618804
- [Result] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Result] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Result] Bruce RA, Kusumi F, Hosmer D. Maximal oxygen intake and nomographic assessment of functional aerobic impairment in cardiovascular disease. Am Heart J. 1973 Apr;85(4):546-62. doi: 10.1016/0002-8703(73)90502-4. No abstract available. PMID 4632004
- [Result] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Result] Campbell-Sills L, Stein MB. Psychometric analysis and refinement of the Connor-davidson Resilience Scale (CD-RISC): Validation of a 10-item measure of resilience. J Trauma Stress. 2007 Dec;20(6):1019-28. doi: 10.1002/jts.20271. PMID 18157881
- [Result] Carver CS. You want to measure coping but your protocol's too long: consider the brief COPE. Int J Behav Med. 1997;4(1):92-100. doi: 10.1207/s15327558ijbm0401_6. PMID 16250744
- [Result] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Result] Fernandez-Berrocal P, Extremera N, Ramos N. Validity and reliability of the Spanish modified version of the Trait Meta-Mood Scale. Psychol Rep. 2004 Jun;94(3 Pt 1):751-5. doi: 10.2466/pr0.94.3.751-755. PMID 15217021
- [Result] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Result] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Result] Herdman M, Badia X, Berra S. [EuroQol-5D: a simple alternative for measuring health-related quality of life in primary care]. Aten Primaria. 2001 Oct 15;28(6):425-30. doi: 10.1016/s0212-6567(01)70406-4. No abstract available. Spanish. PMID 11602124
- [Result] Lyubomirsky, S. and H. S. Lepper (1999).
- [Result] Morán, C., R. Landero, et al. (2009).
- [Result] Munguia-Izquierdo D, Legaz-Arrese A, Mannerkorpi K. Transcultural adaptation and psychometric properties of a Spanish-language version of physical activity instruments for patients with fibromyalgia. Arch Phys Med Rehabil. 2011 Feb;92(2):284-94. doi: 10.1016/j.apmr.2010.10.019. PMID 21272726
- [Result] Munguia-Izquierdo D, Segura-Jimenez V, Camiletti-Moiron D, Alvarez-Gallardo IC, Estevez-Lopez F, Romero A, Chillon P, Carbonell-Baeza A, Ortega FB, Ruiz JR, Delgado-Fernandez M. Spanish adaptation and psychometric properties of the Sedentary Behaviour Questionnaire for fibromyalgia patients: the al-Andalus study. Clin Exp Rheumatol. 2013 Nov-Dec;31(6 Suppl 79):S22-33. Epub 2013 May 27. PMID 23710552
- [Result] Munguia-Izquierdo D, Segura-Jimenez V, Camiletti-Moiron D, Pulido-Martos M, Alvarez-Gallardo IC, Romero A, Aparicio VA, Carbonell-Baeza A, Delgado-Fernandez M. Multidimensional Fatigue Inventory: Spanish adaptation and psychometric properties for fibromyalgia patients. The Al-Andalus study. Clin Exp Rheumatol. 2012 Nov-Dec;30(6 Suppl 74):94-102. Epub 2012 Dec 14. PMID 23261007
- [Result] Notario-Pacheco B, Solera-Martinez M, Serrano-Parra MD, Bartolome-Gutierrez R, Garcia-Campayo J, Martinez-Vizcaino V. Reliability and validity of the Spanish version of the 10-item Connor-Davidson Resilience Scale (10-item CD-RISC) in young adults. Health Qual Life Outcomes. 2011 Aug 5;9:63. doi: 10.1186/1477-7525-9-63. PMID 21819555
- [Result] Panagiotakos DB, Pitsavos C, Stefanadis C. Dietary patterns: a Mediterranean diet score and its relation to clinical and biological markers of cardiovascular disease risk. Nutr Metab Cardiovasc Dis. 2006 Dec;16(8):559-68. doi: 10.1016/j.numecd.2005.08.006. Epub 2006 Feb 9. PMID 17126772
- [Result] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Result] Rikli RE, Jones CJ. Development and validation of criterion-referenced clinically relevant fitness standards for maintaining physical independence in later years. Gerontologist. 2013 Apr;53(2):255-67. doi: 10.1093/geront/gns071. Epub 2012 May 20. PMID 22613940
- [Result] Rodriguez, F. A., N. Gusi, et al. (1998).
- [Result] Rosenberg DE, Norman GJ, Wagner N, Patrick K, Calfas KJ, Sallis JF. Reliability and validity of the Sedentary Behavior Questionnaire (SBQ) for adults. J Phys Act Health. 2010 Nov;7(6):697-705. doi: 10.1123/jpah.7.6.697. PMID 21088299
- [Result] Ruiz-Ruiz J, Mesa JL, Gutierrez A, Castillo MJ. Hand size influences optimal grip span in women but not in men. J Hand Surg Am. 2002 Sep;27(5):897-901. doi: 10.1053/jhsu.2002.34315. PMID 12239682
- [Result] Spielberger CD, Gorsuch RL, et al., Eds. (2002). STAI: Manual del Cuestionario de Ansiedad Estado-Rasgo. Madrid, TEA Ediciones.
- [Result] Spittaels H, Foster C, Oppert JM, Rutter H, Oja P, Sjostrom M, De Bourdeaudhuij I. Assessment of environmental correlates of physical activity: development of a European questionnaire. Int J Behav Nutr Phys Act. 2009 Jul 6;6:39. doi: 10.1186/1479-5868-6-39. PMID 19580645
- [Result] Spittaels H, Verloigne M, Gidlow C, Gloanec J, Titze S, Foster C, Oppert JM, Rutter H, Oja P, Sjostrom M, De Bourdeaudhuij I. Measuring physical activity-related environmental factors: reliability and predictive validity of the European environmental questionnaire ALPHA. Int J Behav Nutr Phys Act. 2010 May 26;7(1):48. doi: 10.1186/1479-5868-7-48. PMID 20504339
- [Result] Vazquez, A. J., R. Jimenez, et al. (2004).
- [Result] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Result] Beck, A. T., R. A. Steer, et al. (2006). BDI-II. Inventario de Depresión de Beck. Buenos Aires, Editorial Paidos.
- [Derived] Marin-Jimenez N, Flor-Alemany M, Ruiz-Montero PJ, Coll-Risco I, Aparicio VA. Effects of concurrent exercise on health-related quality of life in middle-aged women. Climacteric. 2023 Apr;26(2):88-94. doi: 10.1080/13697137.2022.2153032. Epub 2022 Dec 15. PMID 36519287
- [Derived] Coll-Risco I, de la Flor Alemany M, Acosta-Manzano P, Borges-Cosic M, Camiletti-Moiron D, Baena-Garcia L, Aparicio VA. The influence of an exercise program in middle-aged women on dietary habits. The FLAMENCO project. Menopause. 2022 Dec 1;29(12):1416-1422. doi: 10.1097/GME.0000000000002071. Epub 2022 Sep 20. PMID 36126236
- [Derived] Aparicio VA, Flor-Alemany M, Marin-Jimenez N, Coll-Risco I, Aranda P. A 16-week concurrent exercise program improves emotional well-being and emotional distress in middle-aged women: the FLAMENCO project randomized controlled trial. Menopause. 2021 Mar 11;28(7):764-771. doi: 10.1097/GME.0000000000001760. PMID 33739319
- [Derived] Marin-Jimenez N, Ruiz-Montero PJ, De la Flor-Alemany M, Aranda P, Aparicio VA. Association of objectively measured sedentary behavior and physical activity levels with health-related quality of life in middle-aged women: The FLAMENCO project. Menopause. 2020 Apr;27(4):437-443. doi: 10.1097/GME.0000000000001494. PMID 32068685
- [Derived] Aparicio VA, Marin-Jimenez N, Coll-Risco I, de la Flor-Alemany M, Baena-Garcia L, Acosta-Manzano P, Aranda P. Doctor, ask your perimenopausal patient about her physical fitness; association of self-reported physical fitness with cardiometabolic and mental health in perimenopausal women: the FLAMENCO project. Menopause. 2019 Oct;26(10):1146-1153. doi: 10.1097/GME.0000000000001384. PMID 31513090
- [Derived] Carbonell-Baeza A, Soriano-Maldonado A, Gallo FJ, Lopez del Amo MP, Ruiz-Cabello P, Andrade A, Borges-Cosic M, Peces-Rama AR, Spacirova Z, Alvarez-Gallardo IC, Garcia-Mochon L, Segura-Jimenez V, Estevez-Lopez F, Camiletti-Moiron D, Martin-Martin JJ, Aranda P, Delgado-Fernandez M, Aparicio VA. Cost-effectiveness of an exercise intervention program in perimenopausal women: the Fitness League Against MENopause COst (FLAMENCO) randomized controlled trial. BMC Public Health. 2015 Jun 17;15:555. doi: 10.1186/s12889-015-1868-1. PMID 26081934